CLINICAL TRIAL: NCT03262389
Title: Comparison of F-18 FDG PET CT and PET MRI With C-11 Acetate PET CT and PET MRI in the Diagnosis of Active Multiple Myeloma Disease: a Pilot Study
Brief Title: Comparison of F-18 FDG and C-11 Acetate PET in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael C Roarke, MD (Other)
Responsible Party: Sponsor-Investigator, Michael C Roarke, MD, Sponsor-Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-007867
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: positron emission tomography (PET); computerized tomography (CT); Magnetic resonance imaging (MRI); Fludeoxyglucose (F-18 FDG); C-11 acetate
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiple Myeloma Patients (Experimental): Participants will receive 4 different techniques of diagnosis: Fludeoxyglucose (F-18 FDG) PET/MRI, Sodium Acetate (C-11 acetate) PET/CT, C-11 PET/MRI, and F-18 FDG PET/CT. Each participant will receive both PET drugs by both diagnostic techniques and is therefore included in the analysis population for the four reporting groups.
  Interventions: Drug: Fludeoxyglucose PET CT; Drug: Sodium Acetate C11 PET CT; Drug: Fludeoxyglucose PET MRI; Drug: Sodium Acetate C11 PET MRI

INTERVENTIONS:
Drug: Fludeoxyglucose PET CT — Route of administration is intravenous. Dose of each injection will be the standard 5 to 10 millicurie (mCi).
  Other Names: F-18 FDG PET CT
Drug: Sodium Acetate C11 PET CT — Route of administration is intravenous. Dose of each injection will be 10 mCi (370 MBq).
  Other Names: C-11 acetate PET CT
Drug: Fludeoxyglucose PET MRI — Route of administration is intravenous. Dose of each injection will be the standard 5 to 10 millicurie (mCi).
  Other Names: F-18 FDG PET MRI
Drug: Sodium Acetate C11 PET MRI — Route of administration is intravenous. Dose of each injection will be 10 mCi (370 MBq).
  Other Names: C11 PET MRI

SUMMARY:
Investigators are doing this study to determine which of four imaging techniques: Fludeoxyglucose Positron Emission Tomography (18 FDG PET) computerized tomography (CT), 18 FDG PET Magnetic resonance imaging (MRI), C-11 acetate PET CT, and C-11 acetate PET MRI) is the best test for finding sites of active myeloma disease.

DETAILED DESCRIPTION:
Participants who are clinically scheduled to undergo F-18 FDG PET/CT myeloma evaluation will also undergo F-18 FDG PET/MRI, and C-11 acetate PET CT/MRI. On Day 1 of study, participants will undergo F-18 FDG PET/CT-MRI. F-18 FDG radiopharmaceutical is infused intravenously, followed by a 60 minute waiting uptake phase. After 60 minutes, participant will undergo PET/CT imaging for 30 minutes. At 90 minutes, participant will undergo PET/MRI imaging for 30 minutes. On Day 2 of study, participants will undergo C-11 PET/CT-MRI. C-11 radiopharmaceutical is infused intravenously, followed by a 10 minute uptake phase. After 10 minutes, participant will undergo PET/CT imaging for 30 minutes, followed by a 60 minute pause with the participant at rest. At the end of 60 minute pause, the participant is given the second C-11 acetate infusion, followed by a 10 minute waiting uptake phase. After 10 minutes, participant will undergo PET/MRI imaging for 30 minutes. On Day 3, study team member makes a phone call to participant for follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients being staged for multiple myeloma as follows: new diagnosis, high risk smoldering multiple myeloma, relapsed as defined by investigator
* Patients who have undergone standard of care workup
* 300 pounds or less
* Can provide informed consent
* Scheduled for a clinically indicated F-18 FDG PET scan
* English speaking

Exclusion Criteria:

* Pregnant, breast feeding
* Concurrent active non-multiple myeloma malignancy
* Contraindication to PET MRI
* Previous Type I or Type II Diabetes mellitus or a fasting blood glucose >150 mg/dl

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2019-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Roarke, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Myeloma (MM) Patients: New diagnosis, high risk smoldering MM, relapse as defined by investigator. Participants received 4 different techniques of diagnosis: Fludeoxyglucose (F-18 FDG) PET/MRI, Sodium Acetate (C-11 acetate) PET/CT, C-11 PET/MRI, and F-18 FDG PET/CT. Each participant received both PET drugs by both diagnostic techniques and is therefore included in the analysis population for the four reporting groups.
  Fludeoxyglucose: Route of administration was intravenous. Dose of each injection was the standard 5 to 10 millicurie (mCi).
  Sodium Acetate C11: Route of administration was intravenous. Dose of each injection was 10 mCi (370 MBq).
Period: Overall Study
Arm/Group | Multiple Myeloma (MM) Patients
Started | 10
Completed | 7
Not Completed | 3
Not completed — Machine malfunction Day 1, no return Day 2 | 1
Not completed — opted out of the study once his clinical FDG PET CT was done. | 1
Not completed — opted out of PET/MR | 1

BASELINE CHARACTERISTICS:
Arm/Group | Multiple Myeloma (MM) Patients
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Black or African American | 1
  Hispanic or Latino | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Multiple Myeloma Lesions Detected
Description: The number of lesions detected in the scans will be averaged for each technique. Two techniques (scans) will be tested on Day 1 and two techniques (scans) will be tested on Day 2.
Time Frame: Day 1, Day 2
Population: Each participant received both PET drugs by both diagnostic techniques (scans) and is therefore included in the analysis population for the four reporting groups.
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Multiple Myeloma (MM) Patients
Number analyzed (Participants) | 7
number of lesions
  C-11 acetate PET CT | 4.6 (5.1)
  C-11 acetate PET MRI | 4.4 (5.2)
  18 FDG PET CT | 1.1 (1.7)
  18 FDG PET MRI | 1.0 (1.8)

2. Secondary Outcome: Visual Image Analysis of Detected Multiple Myeloma Lesions
Description: The visual image analysis scale has a range of 0-4: (0 no uptake; 1 benign, 2 probably benign, 3 probably malignant, 4 malignant).
Time Frame: Approximately one month after Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multiple Myeloma (MM) Patients
Number analyzed (Participants) | 7
score on a scale
  C-11 acetate PET CT | 3.1 (1.9)
  C-11 acetate PET MRI | 3.3 (1.8)
  18 FDG PET CT | 1.9 (2.0)
  18 FDG PET MRI | 2.0 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to one day following the last administration of study treatment, for at total of approximately 3 days.
Arm/Group | Multiple Myeloma (MM) Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03262389/Prot_SAP_000.pdf